CLINICAL TRIAL: NCT02602886
Title: Exposure and Response Prevention Therapy for Obsessive-compulsive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Shanghai Hongkou Mental Health Center (Unknown); West China Hospital (Other); Suzhou Guangji Hospital (Unknown); First Affiliated Hospital of Xinjiang Medical University (Other); The SHSMU-ION Research Center for Brain Disorders (Unknown)
Responsible Party: Principal Investigator, Bomin Sun, Director of Functional Neurosurgery Department, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCD#020
Record Dates: First submitted 2015-11-05; First posted 2015-11-11 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exposure and Response Prevention Therapy (Experimental)
  Interventions: Behavioral: Exposure and Response Prevention Therapy

INTERVENTIONS:
Behavioral: Exposure and Response Prevention Therapy — The treatment includes both therapist-supervised and self-controlled exposure and ritual prevention exercises. 2 sessions per week, up to 15 sessions in total. Session time is 90 minutes. The majority of in-session time is spent conducting in vivo exposures. When engaging in E/RP tasks, patients are instructed to refrain from ritual engagement. Between-session homework is given the patient practicing the within-session E/RP task up to 90 minutes each day. Clinicians supplement E/RP with other cognitive-behavioral interventions including motivational strategies for resistant patients, Socratic dialogue, and behavioral experiments to test the validity of erroneous cognitions.

SUMMARY:
The purpose of this research study is to evaluate whether Exposure and Response Prevention Therapy (ERP) can help adults with obsessive-compulsive disorder (OCD) in China following a training of professionals and ongoing consultation.

DETAILED DESCRIPTION:
The purpose of this research study is to evaluate whether Exposure and Response Prevention Therapy (ERP) can help adults with obsessive-compulsive disorder (OCD) in China following a training of professionals and ongoing consultation.The treatment time for each participant is approximately 12 weeks. This includes the time between the referral and the beginning of treatment, the treatment sessions, and the 1-month follow-up time. Therapy sessions will take place twice per week for 15 sessions total and last about 90 minutes each. In addition to the therapy sessions, participants will have 3 separate assessments. These assessments will occur (1) right after they agree to participate in the study, (2) immediately after ERP ends, and (3) 1 month after ERP ends. The assessments will take about 1 ½ hours each.

ELIGIBILITY:
Inclusion Criteria:

* Minimum score of >16 on the Y-BOCS; this score indicates clinically significant OCD symptom severity;
* Medically healthy
* Outpatient men and women age 18 years and older;
* Meets DSM-IV criteria for a diagnosis of OCD as determined by the MINI. OCD is the primary psychiatric diagnosis (i.e., it is defined by the patient as the most important source of current distress);
* Able to communicate meaningfully with the investigators and competent to provide written informed consent. IQ estimate > 85 standard score.

Exclusion Criteria:

* Current clinically significant suicidality or individuals who have engaged in suicidal behaviors within the past 12 months will be excluded and referred for appropriate clinical intervention;
* Presence of any clinical features requiring a higher level of care (inpatient or partial hospital treatment);
* Current or past DSM-IV bipolar disorder (Current or past unipolar depression is not an exclusion criterion. We will allow comorbid depression, to ensure that we are treating a representative OCD sample. Depression is the most common complication in OCD, and about one third of the OCD clinical samples are depressed.)
* Schizophrenia, schizoaffective disorder, or any other current or lifetime DSM-IV psychotic disorder;
* Current or recent (within 3 months of study entry) DSM-V alcohol or drug dependence or abuse (other than nicotine), or a positive urine drug screen for any illicit substances of abuse;
* Estimated IQ <85 on the WASI, mental retardation, dementia, brain damage, or other cognitive impairment that would interfere with the capacity to participate in the study and complete self-report measures;
* Any medical conditions that might contraindicate use of the study treatments, as determined by medical physical and laboratory tests by the study physicians;
* Presence of any significant and/or unstable medical illness which might lead to hospitalization during the study duration; subjects with a stable medical condition may participate with the agreement of the subject's physician and the study physician who performs the study physical exam;
* Concurrent psychotherapy of any type (e.g., CBT/ERP, supportive, psychodynamic) and duration;
* History of adequately-delivered exposure-based cognitive-behavioral therapy (i.e., 10 or more sessions of specific and regular exposure and/or response prevention assignments; as needed and with patients' written permission we will confer with prior treatment providers).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in Yale-Brown Obsessive Compulsive Scale (Y-BOCS) Score | Baseline, upon ERP completion(average 7.5 weeks), 1 month after ERP completion

SECONDARY OUTCOMES:
Change in Florida Obsessive-Compulsive Inventory (FOCI) Score | Baseline, after every session(average 3.5 days), upon ERP completion(average 7.5 weeks), 1 month after ERP completion
Change in Obsessive-Compulsive Inventory-Revised (OCI-R) Score | Baseline, upon ERP completion(average 7.5 weeks), 1 month after ERP completion
Change in Hamilton Anxiety Scale, Hamilton Depression Scale-17 Score | Baseline, upon ERP completion(average 7.5 weeks), 1 month after ERP completion
Change in Obsessional beliefs questionnaire (OBQ-44) Score | Baseline, upon ERP completion(average 7.5 weeks), 1 month after ERP completion
Change in Patient EX/RP Adherence Scale (PEAS) Score | From the fourth session(average 1.5 weeks), upon ERP completion(average 7.5 weeks), 1 month after ERP completion
Disability: Change in Sheehan Disability Scale | Baseline, upon ERP completion(average 7.5 weeks), 1 month after ERP completion
Disability: Change in WHO disability assessment 2.0 | Baseline, upon ERP completion(average 7.5 weeks), 1 month after ERP completion
Treatment Ambivalence Questionnaire (TAQ) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bomin Sun, MD, PhD, Study Director — Ruijin Hospital
Locations (5):
- China (5):
  - Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Chengdu, Sichuan
  - Shanghai Hongkou Mental Health Center, Shanghai Shi
  - Suzhou Guangji Hospital, Suzhou
  - The First Hospital affiliated to XinJiang Medical University, Ürümqi

IPD SHARING:
Plan to Share IPD: No